CLINICAL TRIAL: NCT05446051
Title: Development and Testing of a Telephone Triage Decision Support System (TTDSS) for Cancer Patients
Brief Title: Development and Testing of a TTDSS for Cancer Patients
Acronym: TTDSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STM-IRB-22B-001
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-08

CONDITIONS: Treatment Side Effects
Keywords: Telephone Triage Decision Support System; Treatment Induced Adverse Events

STUDY DESIGN:
Intervention Model Description: Experimental Group：New patients and take the TRAEs Questionnaire on week. Control Group：Old patients and usual care.
Who Masked: Participant
Masking Description: Single-blind(Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): New patients and take the TRAEs Questionnaire on week.
  Interventions: Device: the Mandarin Version of the electronic patient self-Reporting of Adverse-events (eRAPID-MV); Device: the telephone triage decision support system (TTDSS)
- Control group (No Intervention): Control Group：Old patients and usual care.

INTERVENTIONS:
Device: the Mandarin Version of the electronic patient self-Reporting of Adverse-events (eRAPID-MV) — Phase I Interventions：eRAPID-MV(TRAEs survey)
  Arms: Experimental Group
Device: the telephone triage decision support system (TTDSS) — Phase I Interventions：TTDSS
  Arms: Experimental Group

SUMMARY:
This study aimed at testing the technical and clinical feasibility of the Mandarin Version of the electronic patient self-Reporting of Adverseev ents (eRAPID-MV) and the telephone triage decision support system (TTDSS) by testing them on patients with breast and colorectal cancer. The hypothesis of this study was the patients with breast and colorectal cancer who received eRAPID-MV and TTDSS were performing better on patient care outcomes and telephone screening service outcomes than patients who had not received eRAPID-MV and TTDSS. A non-randomized comparison trial was performed in St. Martin De Porres Hospital, Taiwan from July 2022 to April 2023. This study employed a quasi-experimental design to collect data from a treatment induced adverse events (TRAEs) questionnaire, a satisfaction questionnaire, and an interview with patients. It used the system usability scale (SUS) to assess data usability. 136 patients with breast cancer or colorectal cancer were unrolled and distributed in two groups. In Phase I, participants were selected based on convenience sampling and non-randomly assigned to an experimental group (N=68). They received chemotherapy and completed the eRAPID-MV measures-based TRAEs survey every week. The control group (N = 68) received usual care. The program duration was 24 weeks. At the end of the program, the researcher recruited participants from the experimental group based on voluntary recruitment for a single interview to assess their views on the eRAPID-MV system. The interview duration was approximately 20-30 minutes. Both groups completed the pre-test and post-test TRAEs questionnaire. In Phase II, when the TRAEs survey indicated a red light for experimental group, the eRAPID-MV system provided automatic recommendations to the patient to seek emergency medical services, or the patient contacted the case manager to deal with severe TRAEs. Simultaneously, the oncology case manager or oncologist received an alarm reminder immediately. Based on the TRAEs survey indication (red or yellow light) and consultation with the patient via a phone call, the oncology case manager reassessed the patient's TRAEs using TTDSS and scheduled their follow-up appointment accordingly. After 72 hours of intervention in Phase II (TTDSS), the first post-test was performed to assess the immediate effects. The long-term effects were evaluated at the end of the intervention, which lasted 180 days (6 months).

DETAILED DESCRIPTION:
This study aimed to understand the use of different educational models (eRAPID-MV) and self-management behaviors of cancer patients in managing treatment-induced side effects at home. To this end, interventions were provided through a decision support system involving telephone triage. Finally, the study explored the effectiveness of the intervention method (eRAPID-MV & TTDSS) on patient care outcomes and telephone triage service outcomes.

Study design/setting This was a prospective, nonrandomized clinical study.Study procedures and data collection were carried out at the outpatient department of St. Martin De Porres Hospital, Taiwan. The trial followed the Declaration of Helsinki and Good Clinical Practice guidelines for trial conduct. Participants a breast surgeon or colorectal surgeon or hematologist oncologist were invited or referred to participate in the research project. Participants provided their written informed consent prior to taking part in this 24-week program. Participants has received a weekly reminder from the APP or emails to complete an online TRAEs (eRAPID-MV) assessment at home. Participants used an electronic device (e.g., smart phone, tablet, computer) with real-time electronic data transfer to the Health Care Information System (HIS). During the study period, participants were compared to a usual care control group on patient care outcomes and telephone screening service outcomes.

Interventions Two key intervention components were standardized across participating hospitals: Phase I Interventions: eRAPID-MV system-a) TRAEs surveys, b) survey feedback reports, and c) patient self-management and clinical alerts; Phase II Interventions: TTDSS.

The Phase I intervention details are as follows: (1) The patients completed the TRAEs survey-18 items. Based on the survey results, the eRAPID-MV system provided a summary report of the traffic signal and recommendations to the patient for seeking medical advice (red or yellow light), and a link to the TRAEs websites for self-management (green light). The TRAEs websites on health education summarized available information from symptom management guidelines, telephone triage protocols for nurses, and published articles. (2) The survey results were also integrated into the hospital information system (HIS) and case management system (Cancer Patient Registry) to enable the clinician and case managers to access report summaries and review patient-reported outcomes for severe TRAEs. (3) All the patients (experimental group) completed the TRAEs survey every week during their active treatment period, and the eRAPID-MV system's automatic schedule was sent to them. (4) The intervention duration was 24 weeks. (5) Participants were asked to fill out a satisfaction survey on weeks 2, 12, and 24. The system usability scale (SUS) was also used on the day of the final survey. Finally, patients were recruited to attend a single interview that assessed their views on the eRAPID-MV system. Participation was voluntary, and the interview lasted approximately 20-30 minutes.

The Phase II intervention details are as follows: (1) a phone consultation with the oncology case manager was determined based on the patient's TRAEs (red or yellow light-experimental group or the need for a return visit). The oncology case manager referred to the last TRAEs data and inquired about the patient's present condition. Based on the information and the purpose of the patient's call, the oncology case manager evaluated the severity of TRAEs by referring to the guidelines for TTDSS. The patient received the best possible recommendation to help manage TRAEs based on a summary report of the traffic signal. When the light was red or yellow, the oncology case manager arranged for immediate outpatient or emergency medical treatment and assisted in hospitalization if necessary. (2) Following Phase II intervention (TTDSS) for 72 hours, the first post-test was performed to assess the immediate effects on the patient. (3) Long-term effects were also evaluated, including the effectiveness of patient care outcomes and telephone triage service outcomes on cancer patients after 24 weeks of intervention. (4) Finally, the oncology case manager asked to attend a single interview that assessed their views on the TTDSS. Participation was voluntary, and the interview lasted approximately 20-30 minutes.

Data collection and management For the 24-week study period, participants were evaluated at baseline, and every week (experimental group) or every 3 weeks (control group) by TRAEs assessment. Participants were asked to complete 3, brief, self-administered questionnaires: the treatment-induced adverse events (TRAEs) questionnaire, satisfaction questionnaire, system usability scale (SUS), and interview with patients (experimental group). All questionnaires and the consent form were translated into Chinese (Traditional) by a certified translator. The TRAEs data were fully integrated into HIS and the case management system (including the Cancer Patient Registry) of St Martin De Porres Hospital (id: STM-IRB-22B-001-2022-04). Data were processed anonymously; therefore, data for which participants' identities could be identified were omitted. Strict safety and confidentiality measures were established in the archives of clinical trial institutions. Every six months, the Institutional Review Board (IRB) will be responsible for checking the status of the study and the quality of the data collected.

Sample size calculation The multiple linear regression statistical method was followed to estimate the sample size of the cluster, and the number of patients required for the study was determined accordingly. The total sample size required for the computer software calculation was 114. Considering the attrition rate of approximately 20%, the estimated sample size for this study was at least 136, and the average sample size for each group was at least 68.

Statistical analysis Descriptive statistics, including means, standard deviations, frequencies, and percentages, and chi-square tests and independent t-tests, were used to test the homogeneity of context-level factors (e.g. demographic characteristics, disease status, and family caregiver support) between the two groups. Binary logistic regression and polynomial linear regression were used to analyze the factors influencing self-management behaviors. Inferential statistics, including paired sample t-test, 2-group sample t-test, Mc Nemar's test, and analysis of covariance (ANCOVA), were used. Following the eRAPID- MV and TTDSS intervention, analyses were performed to assess changes in patient care outcomes (TRAEs severity, disconnection rate, hospitalization rate, retention rate, and completion rate) and triage service outcomes (ease of use of the system).

ELIGIBILITY:
Inclusion Criteria:

* Are age 20 years or over
* Aare eligible diagnosed with ICD-10 colorectal cancer (C18-C21) or breast cancer (C50),
* Received chemotherapy for at least three months were Chinese literate.

Exclusion Criteria:

* Classification 0 (diagnosed in one hospital, treated in other hospitals) and category 3 (diagnosed in other hospitals, treated in other hospitals) cases of cancer
* deceased patients
* patients without a local telephone, mobile phone, or Internet access at home
* illiterate patients or patients who cannot use mobile phones or the Internet.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-11-06 (Estimated); Study Completion 2024-04-06 (Estimated)

PRIMARY OUTCOMES:
TRAEs severity | 24 weeks
  Operational definitions:
  Calvett et al. (2021) and Richards et al. (2020) were used to develop the item assessment and severity grading of TRAEs based on the version 5.0 CTCAE scale (visualization of red, yellow, and green lights). Green events (CTCAE-1): mild AEs with self-management advice only; yellow events (CTCAE-2): moderate AEs with self-management advice, and recommend patient to a phone consultation with the oncology case manager; Red events (CTCAE-Grade 3 and 4): Severe AE recommend patients to be referred to a hospital as soon as possible within 24 hours. TRAEs severity was then graded on a scale of 1-4, with 4 being the most severed and 1 being not severed at all.
loss to follow-up rate | 24 weeks
  Operational definition:
  The loss to follow-up rate is defined according to accreditation of Cancer Care Program by the Taiwan Cooperative Oncology Group. The numerator is the number of missing cases for breast and colorectal cancers for 3 months; the denominator is the number of missing cases for breast and colorectal cancers (total number of cases - number of deaths).
hospitalization rates | 24 weeks
  Operational definition:
  TRAEs with a severity rating of yellow events and red events that require further hospitalization after assessment by an outpatient or emergency clinician. The numerator is the actual number of hospitalizations in the denominator; the denominator is the total number of severe yellow events and red events of TRAEs (excluding the number of deaths).
Retention rate | 24 weeks
  Operational definition:
  The retention rate is defined according to accreditation of Cancer Care Program by the Taiwan Cooperative Oncology Group. The numerator is the number of missing cases for breast and colorectal cancers for 6 months; The denominator is the number of new cases of breast cancer and colorectal cancer (Class 1~2) diagnosed in the hospital during the year.
treatment completion rates | 24 weeks
  Operational definition:
  The treatment completion rate is defined according to accreditation of Cancer Care Program by the Taiwan Cooperative Oncology Group. The numerator is the number of cases in the denominator in which a single type of treatment (e.g. chemotherapy, radiation therapy) was completed within 6 months of the first treatment.; The denominator is the number of cases of breast cancer and colorectal cancer newly diagnosed (Class 1~2) and treated (surgery, chemotherapy, radiotherapy) in our hospital in the current year.

SECONDARY OUTCOMES:
compliance with care recommendations | 24 weeks
  Operational definition:
  The compliance scale was measured by the researcher's self-developed the compliance with care recommendations based on the TTDSS with a dichotomous scale of compliance (1) and non-compliance (0), with a score range of 0-1, the higher scores representing higher compliance.
patient satisfaction | 24 weeks
  Operational definition:
  The satisfaction scales of eRAPID-MV and TTDSS were self-developed by the investigator with reference to relevant literature; one question each on this scale was measured on a five-point scale, "very dissatisfied" (1 point), "satisfied" (2 points), "fair" (3 points), "satisfied" (4 points), and "very satisfied" (5 points), with scores ranging from 1 to 5, with higher scores indicating higher levels of patient satisfaction.
system usability | 24 weeks
  Operational definition:
  Originally the System Usability Scale (SUS) created by John Brooke in 1986. SUS provides a quick and reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree (5 point) to Strongly disagree (1 point). The score range is 0-100, and the higher the score, the higher the usability of the system. In order to increase the reliability of the questionnaire, the odd numbered questions were used as positive questions and the even numbered questions were used as negative questions, and the survey was conducted in a positive and negative crossover manner.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Ping Liu, Director, Study Chair — Ministry of Health and Welfare
Locations (1):
- St. Martin De Porres Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No